CLINICAL TRIAL: NCT00519116
Title: An Open-label, Concentration-controlled, Randomized, 6-month Study of 'Standard Dose' Tacrolimus + Sirolimus + Corticosteroids Compared to 'Reduced-dose' Tacrolimus + Sirolimus + Corticosteroids in Renal Allograft Recipients
Brief Title: Study Comparing Standard Dose and Reduced Dose Tacrolimus With Sirolimus in Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468E1-100539
Record Dates: First submitted 2007-07-27; First posted 2007-08-21 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Sirolimus; Tacrolimus

INTERVENTIONS:
Drug: Rapamune® (Sirolimus)
Drug: Tacrolimus
Drug: Perioperative Corticosteroids — The corticosteroids use was left up to the investigators decision.

SUMMARY:
The study evaluated renal graft function (based on the calculated creatinine clearance) 6 months after kidney transplantation in patients receiving either a regimen of 'reduced-dose' tacrolimus + sirolimus + corticosteroids or a regimen of 'standard-dose' tacrolimus + sirolimus + corticosteroids.

DETAILED DESCRIPTION:
The study evaluated renal graft function (based on the calculated creatinine clearance) 6 months after kidney transplantation in patients receiving either a regimen of 'reduced-dose' tacrolimus + sirolimus + corticosteroids or a regimen of 'standard-dose' tacrolimus + sirolimus + corticosteroids. The two treatment groups were also compared with respect to the incidence of acute graft rejection at 6 months and patient and graft survival at 6 months after transplantation.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age
* End-stage renal disease in patients receiving a primary or secondary renal allograft from a cadaveric, living-unrelated, or living-related mismatched donor
* Patients with a secondary transplant must have maintained a primary graft for at least 6 months

Exclusion criteria:

* Planned antibody induction
* Multiple organ transplants
* History of malignancy within five years of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2000-10; Study Completion 2001-08

PRIMARY OUTCOMES:
Calculated creatinine clearance at month 6 post transplantation | 6 months

SECONDARY OUTCOMES:
Patient and graft survival at 6 months post transplantation; the safety of sirolimus + corticosteroids given concomitantly with reduced or standard dose tacrolimus | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer